CLINICAL TRIAL: NCT07236710
Title: Evolving Strategies in Placenta Accreta Spectrum Management: A Ten-Year Institutional Review
Brief Title: Observation of Strategies in Placenta Accreta Spectrum Management
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ayman Saad zaghlol Abdallah, Resident doctor, Assiut University
Other Study IDs: placenta Accreta management
Record Dates: First submitted 2025-11-15; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Placenta Accreta Management

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
• Placenta accreta spectrum (PAS) disorders represent a significant obstetric challenge, characterized by abnormal adherence of the placenta to the uterine wall, leading to potentially life-threatening hemorrhage (ACOG 2020; RCOG 2018; Jauniaux 2019) during delivery. PAS includes placenta accreta (attachment to the myometrium), increta (invasion into the myometrium), and percreta (penetration through the uterine serosa, often involving adjacent organs). The incidence of PAS is rising globally, largely attributed to the increased rates of cesarean section and uterine surgeries (Bowman 2021).

Effective management of PAS is crucial to prevent severe maternal morbidity and mortality. The cornerstone of management remains surgical intervention, with cesarean hysterectomy being the traditional gold standard (Eller 2009; ACOG 2020), especially in cases of extensive invasion. However, conservative and fertility-preserving surgical techniques have emerged in recent years as viable alternatives in selected cases (Jauniaux 2019).

In Assiut university hospital, diverse surgical approaches are practiced depending on the extent of placental invasion, surgeons expertise, and patient fertility desires. These include cesarean hysterectomy, segmental uterine resection, the Triple-P procedure, and uterus-preserving methods such as leaving the placenta in situ. (ijrcog) A notable contribution to conservative PAS management in Egypt is the Placental Pouch Closure technique. This technique involves careful resection of the invaded uterine wall followed by multilayered closure of the resulting myometrial defect (the "placental pouch"), thereby controlling hemorrhage while preserving uterine integrity.

(Zahran et al. 2020) .

• This retrospective study aims to evaluate the pattern and outcomes of various surgical approaches used in the management of placenta accreta spectrum disorders over a 10-year period at a Assiut university hospital. Special attention will be paid to the adoption, safety, and effectiveness of conservative techniques

ELIGIBILITY:
Inclusion Criteria:

* - Women diagnosed with PAS (accreta, increta, percreta).
* Deliveries conducted at Women's Health Hospital.
* Age 18-50 years.
* Availability of complete medical records and operative details.

Exclusion Criteria:

* - Patients with incomplete records or missing surgical reports.
* Cases managed outside the hospital.

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — All pregnant women diagnosed with placenta accreta spectrum disorders during the study period
Study Population: All pregnant women diagnosed with placenta accreta spectrum disorders during the study period
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2027-10-20 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Patterns of management over time | 10 years
  Patterns of management of placenta Accreta in retrospective way on the last 10 years

REFERENCES:
- [Result] Eller AG, Porter TF, Soisson P, Silver RM. Optimal management strategies for placenta accreta. BJOG. 2009 Apr;116(5):648-54. doi: 10.1111/j.1471-0528.2008.02037.x. Epub 2009 Feb 4. PMID 19191778
- [Result] Jauniaux E, Ayres-de-Campos D, Langhoff-Roos J, Fox KA, Collins S; FIGO Placenta Accreta Diagnosis and Management Expert Consensus Panel. FIGO classification for the clinical diagnosis of placenta accreta spectrum disorders. Int J Gynaecol Obstet. 2019 Jul;146(1):20-24. doi: 10.1002/ijgo.12761. PMID 31173360
- [Result] Jauniaux E, Alfirevic Z, Bhide AG, Belfort MA, Burton GJ, Collins SL, Dornan S, Jurkovic D, Kayem G, Kingdom J, Silver R, Sentilhes L; Royal College of Obstetricians and Gynaecologists. Placenta Praevia and Placenta Accreta: Diagnosis and Management: Green-top Guideline No. 27a. BJOG. 2019 Jan;126(1):e1-e48. doi: 10.1111/1471-0528.15306. Epub 2018 Sep 27. No abstract available. PMID 30260097